CLINICAL TRIAL: NCT01412268
Title: Study of Eating Habits and Addiction Changes in Short and Long Time Follow-up in Morbidly Obese Patients Who Undergo Bariatric Surgery.
Brief Title: Does Bariatric Surgery Changes Eating Habits and Addiction in Morbid Obesity?
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Suleyman Bozkurt, Associated Professor, Bezmialem Vakif University
Other Study IDs: BAVUGC-1
Record Dates: First submitted 2011-08-08; First posted 2011-08-09 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Obesity
Keywords: Obesity; Bariatric surgery; Behavioral changes; Eating habits; Eating addiction
MeSH Terms: conditions — Obesity; Feeding Behavior

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
1. Obesity is a big health problem worldwide.
2. Mostly obese people have food addiction and bad eating habits.
3. Bariatric surgery is a good alternative for patients who failed to loose weight with other measures like behavioral changes, activities and sports, diet, etc..
4. The investigators know the changes occurred after surgery in eating habits due to restrictive and malabsorptive feature of the surgery performed.
5. There is no study in the literature to measure these changes.
6. The investigators will try to detect these kind of behavioral changes by a survey before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with BMI > 40 kg/m2
* Patients with BMI > 35 kg7m2 < 40 kg/m2 but with comorbidity
* Patients > 18 years old
* Patients who sign the inform consent
* Patients who have no psychiatric disease
* Patients who have no endocrine disorders

Exclusion Criteria:

* All obese patients who do not fulfill the criteria above mentioned

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with BMI > 40 kg/m2 Patients with BMI > 35 kg7m2 < 40 kg/m2 but with comorbidity Patients > 18 years old Patients who sign the inform consent Patients who have no psychiatric disease Patients who have no endocrine disorders
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Actual)

REFERENCES:
- [Derived] Sevincer GM, Konuk N, Bozkurt S, Coskun H. Food addiction and the outcome of bariatric surgery at 1-year: Prospective observational study. Psychiatry Res. 2016 Oct 30;244:159-64. doi: 10.1016/j.psychres.2016.07.022. Epub 2016 Jul 12. PMID 27479107